CLINICAL TRIAL: NCT06041763
Title: Outcomes Following Meniscal Repair With the BEAR Implant: A Randomized Controlled Trial
Brief Title: Bridge-Enhanced ACL Repair (BEAR) in Meniscus Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-00813
Record Dates: First submitted 2023-09-12; First posted 2023-09-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Meniscus Tear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BEAR Implant (Experimental): Adult patients with meniscus injury indicated for isolated meniscus repair. In the experimental group, the BEAR Implant will be utilized in the repair procedure.
  Interventions: Procedure: Meniscal Repair Procedure; Device: BEAR Implant
- Standard Repair (Active Comparator): adult patients with meniscus injury indicated for isolated meniscus repair. In the standard repair group, participants will undergo an isolated meniscus repair without the implant.
  Interventions: Procedure: Meniscal Repair Procedure

INTERVENTIONS:
Procedure: Meniscal Repair Procedure — All meniscal repairs will be performed by the surgeons who are listed as investigators for the study. Meniscal repair consists of arthroscopic suturing of torn fragments. This takes approximately 20 minutes. In the interventional group, the BEAR implant will be inserted through preexistent arthroscopic portals after repair is complete. This will take an additional 2 minutes.
Device: BEAR Implant — The BEAR Implant (22 mm in diameter and 45mm in length) is cylindrical in shape and comprised of collagen and extracellular matrix derived from bovine connective tissue, which has been cleaned, disinfected and processed by a proprietary manufacturing method. The implant has been terminally sterilized by electron-beam inadiation and is intended to be used with up to 10 ml of autologous blood drawn during the surgical implantation procedure. The BEAR Implant is resorbed within 8 weeks and replaced with a fibrovascular repair tissue.
  Arms: BEAR Implant

SUMMARY:
The bridge-enhanced ACL repair (BEAR) implant is a collagen-based scaffold loaded with whole blood. It is designed to promote healing in the setting of intraarticular knee pathology. This study would compare clinical outcomes and synovial fluid cytokine profiles in patients who undergo isolated meniscal repair with or without the BEAR implant.

ELIGIBILITY:
Inclusion Criteria:

• History of meniscus injury indicated for isolated repair, without concomitant ligament reconstruction or repair, cartilage repair procedure, or osteotomy.

Exclusion Criteria:

* Patients who are undergoing meniscal repair for displaced bucket-handle meniscal tears
* Patients with a history of blood-borne diseases including HIV, hepatitis B virus, hepatitis C virus, human T-lymphotropic virus, and syphilis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in International Knee Documentation Committee (IKDC) Subjective Knee Form Score | Baseline, 1 Year Post-Procedure
  10-item assessment of knee-related symptoms at the present moment and over the previous 4 weeks. Each item is rated according to presence of symptoms. The raw score is the sum of responses and is rescaled to a total score ranging from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Change in Lysholm Scale Score | Baseline, 1 Year Post-Procedure
  8-item assessment of knee-related activity and problems at the present moment. Each item is rated on a Likert-type scale. The total score is the sum of responses and ranges from 0 to 100, with higher scores indicating greater level of function/lower level of symptoms.
Change in Visual Analogue Scale (VAS) Score | Baseline, 1 Year Post-Procedure
  One-item assessment of pain on the current day. Pain is rated on a scale from 0 (no pain) to 10 (worst possible, unbearable, excruciating pain); the total score is the numerical rating.
Incidence of Repair Failure | Up to 1 Year Post-Procedure
  Instances of failure of the meniscal repair.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Gonzalez-Lomas, MD Gonzalez-Lomas, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: isabel.wolfe@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to isabel.wolfe@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.